CLINICAL TRIAL: NCT05741697
Title: High Flow Nasal Cannula Versus Non-invasive Ventilation in Managing Acute Exacerbation of Bronchiectasis Patients
Brief Title: HFNC in Management of Bronchiectasis Exacerbation
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: WGEKHALEEL (Unknown); AARMHUSSIEN (Unknown)
Responsible Party: Principal Investigator, Ahmad Shaddad, lecturer of pulmonology, Assiut University
Other Study IDs: 2627378373
Record Dates: First submitted 2023-02-12; First posted 2023-02-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient need NIV ventillation: Patients will be eligible for enrolment if they are diagnosed with bronchiectasis and admitted to the respiratory intensive care unit (RICU); requiring ventilator support without invasive mechanical ventilation and will need NIV
  Interventions: Drug: bi-level ventillation
- patient need HFNC: Patients will be eligible for enrolment if they are diagnosed with bronchiectasis and admitted to the respiratory intensive care unit (RICU); requiring ventilator support without invasive mechanical ventilation and will need HFNC

INTERVENTIONS:
Drug: bi-level ventillation — non-invasive mechanical ventilation
  Other Names: HFNC
  Groups: Patient need NIV ventillation

SUMMARY:
Patients with Bronchiectasis experience exacerbations with hypercapnic respiratory failure associated with an increased respiratory workload that may require intensive care unit (ICU) admission due to the inability of the respiratory muscles to compensate for increased demand. These exacerbations are frequently treated with noninvasive ventilation (NIV).

DETAILED DESCRIPTION:
NIV has been shown to unload the respiratory muscles, increase alveolar ventilation and gas exchange and reverse the rapid and shallow breathing pattern commonly adopted by bronchiectasis patients with advanced lung disease.

NIV is a cornerstone therapy for hypercapnic acute respiratory failure. Still, there is also an increasing interest in high-flow nasal cannula (HFNC) as a potential alternative treatment in this indication. HFNC delivers an actively heated and fully humidified gas mixture with flow rates up to 60 L/min and adjustable FiO2 from 21 to 100%. The high flow rates generate small amounts of positive end-expiratory pressure (PEEP) that may help counterbalance the effects of intrinsic PEEP (PEEPi) on the work of breathing and might act by washing out of the physiological dead space. Furthermore, it could help to facilitate secretion clearance from the humidified gas.

Studies have demonstrated the benefits of HFNC in acute hypoxemic respiratory failure, after cardiothoracic surgery, and in preventing post-extubation failure among unselected cohorts of critically ill patients during weaning from invasive mechanical ventilation.

However, the current evidence of using HFNC in patients with hypercapnic acute respiratory failure is limited. We aime to spotlight this research area.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for enrolment if diagnosed with bronchiectasis and admitted to the respiratory intensive care unit (RICU), requiring ventilator support without invasive mechanical ventilation.

Exclusion Criteria:

* Age: less than 18 years. Patients with post-arrest encephalopathy. Patient with the previous tracheotomy. Patients who received invasive ventilatory support. Patients with end-organ failure.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be eligible for enrolment if diagnosed with bronchiectasis and admitted to the respiratory intensive care unit (RICU), requiring ventilator support without invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy and patient compliance of high flow nasal canula system in comparison to Noninvasive mechanical ventilation in management of acute exacerbation of Bronchiectasis | March 2023 to December 2023
  The duration of ICU admission days and the patient compliance to both devices will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Shaddad, Principal Investigator — Assiut University
Locations (1):
- Assiut University-Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No